CLINICAL TRIAL: NCT00493766
Title: A Phase IA/IB, Two Arm, Multi-center, Open-label, Dose Escalation Study of Oral LBH589 Alone and in Combination With IV Docetaxel and Oral Prednisone in Hormone Refractory Prostate Cancer (HRPC)
Brief Title: Safety of LBH589 Alone and in Combination With IV Docetaxel and Prednisone
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Because of a strategic decision by Novartis
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CLBH589B2105
Record Dates: First submitted 2007-06-26; First posted 2007-06-28 (Estimated); Last update posted 2020-12-19 (Actual); Status verified 2012-11

CONDITIONS: Hormone Refractory Prostate Cancer
Keywords: LBH589; Prostate Cancer; HRPC; Hormone Refractory Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Panobinostat

ARMS (2):
- oral LBH589 alone (Experimental)
  Interventions: Drug: LBH589
- oral LBH589 + IV docetaxel + oral prednisone (Experimental)
  Interventions: Drug: LBH589

INTERVENTIONS:
Drug: LBH589

SUMMARY:
This is a parallel, two-arm, open-label, multicenter phase IA/IB study of LBH589 (oral formulation) alone and in combination with docetaxel in patients with progressing hormone refractory prostate cancer. This study is designed to determine the maximum tolerated dose of LBH589 as a single agent and in combination with docetaxel and prednisone 5 mg two times a day , and to characterize the safety, tolerability, biologic activity and pharmacokinetic profile

ELIGIBILITY:
Inclusion criteria:

* Histologically documented adenocarcinoma of the prostate.
* Patients must have metastatic disease with at least one measurable soft tissue lesion that can be assessed by computerized tomography (CT), or magnetic resonance imaging (MRI) and/or detectable lesion(s) on bone scintigraphy scan. Patients with only elevated prostate specific antegen (PSA) levels are not eligible for entry.
* Patients who have undergone medical castration must continue Luteinizing hormone-releasing hormone (LHRH) agonist or antagonist therapy during study treatment
* Patients must be able to provide written informed consent

Exclusion criteria:

* Patients with prior or concurrent brain metastases
* Impaired cardiac, gastrointestinal, kidney, or liver function
* Use of therapeutic androgens

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2006-05; Primary Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
• To determine the maximum-tolerated dose (MTD) and dose-limiting toxicity (DLT) of esca-lating doses of LBH589 in adult men with HRPC. | at study start and at study end
• To determine the MTD and DLT of escalating doses of LBH589 in combination with a stan-dard dose of docetaxel q3wks and daily Prednisone® in adult men with HRPC. | at study start and at study end

SECONDARY OUTCOMES:
• To characterize the safety and tolerability of LBH589 alone and in combination with do-cetaxel and Prednisone® including acute and chronic toxicities | at study start and at study end
• To characterize the single-dose and multidose pharmacokinetic (PK) profiles of LBH589 alone and in combination with docetaxel and Prednisone®. To characterize the PK profiles of docetaxel alone and in combination with LBH589. | at study start and at study end

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (5):
- United States (5):
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Washing University School of Medicine, St Louis, Missouri
  - Nevada Cancer Institute, Las Vegas, Nevada
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Duke University Medical Center, Durham, North Carolina

REFERENCES:
- See also: Results for CLBH589B2105 can be found on the Novartis Clinical Trial Results Website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=2939